CLINICAL TRIAL: NCT06018896
Title: Vitamin C to Quality of Life in Patients With Terminal Stage Pancreatic Cancer
Acronym: PTCA199-4
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-4
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Pancreatic Cancer; Terminal Cancer
Keywords: ascorbate; anemia; quality of life; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Anemia | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ascorbate (Experimental): For patients with baseline serum Vitamin C concentration < 65 μmol/L, intravenous Vitamin C 10 g × 7 days, intravenous Vitamin C 4 g × 7 days, intravenous Vitamin C 2 g × 7 days, followed by continuously 900 mg/day, three times a day, orally. For patients with baseline serum Vitamin C concentration ≥ 65 μmol/L, continuously 900 mg/day, three times a day, orally.
  Interventions: Drug: Ascorbate

INTERVENTIONS:
Drug: Ascorbate — For patients with baseline serum Vitamin C concentration < 65 μmol/L, intravenous Vitamin C 10 g × 7 days, intravenous Vitamin C 4 g × 7 days, intravenous Vitamin C 2 g × 7 days, followed by continuously 900 mg/day, three times a day, orally. For patients with baseline serum Vitamin C concentration ≥ 65 μmol/L, continuously 900 mg/day, three times a day, orally.
  Other Names: Vitamin C

SUMMARY:
The purpose of this study is to evaluate the efficacy of vitamin C in improving the quality of life for metastatic pancreatic cancer patients who are resistant to chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. In 2011, a trial has shown that oxaliplatin, irinotecan, fluorouracil, and leucovorin (FOLFIRINOX) was associated with a survival advantage but had increased toxicity. In 2013, the Metastatic PAncreatic Cancer Trial (MPACT) has confirmed the efficacy of gemcitabine combined with nab-paclitaxel as the first-line treatment to metastatic pancreatic cancer. However, the side-effects related to chemotherapy including anemia, hand/foot numbness, fatigue, nausea, and malnutrition have impaired the quality of life for patients.

Vitamin C, also called ascorbate, is an essential nutrient for the human body. It modulates metabolism, immune reaction, collagen synthesis, and iron absorption. Some studies have shown that high-dose intravenous Vitamin C may be effective against various types of cancer. Meanwhile, medium or low dose of Vitamin C may increase iron absorption, improve anemia, alleviate pain and hand/foot numbness, and thus improve the quality of life for patients with terminal stage pancreatic cancer.

The purpose of this study is to evaluate the efficacy of vitamin C on improving the quality of life for metastatic pancreatic cancer patients who are resistant to two lines of systemic chemotherapy, including gemcitabine based, fluorouracil based, or other regimen. Twenty patients who have tumor progression after receiving two lines of chemotherapy will be recruited. These patients will receive Vitamin C and the dosage is based on the concentration of baseline serum Vitamin C concentration. Quality of life, rate of hand/foot numbness, severity of pain, rate of anemia, and overall survival are measured every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
* Tumor progression after two lines of chemotherapy.
* Adequate organ performance based on laboratory blood tests.
* Presence of at least of one measurable lesion in agreement to Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
* The expected survival ≥ 1 months.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Active second primary malignancy or history of second primary malignancy.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Pregnant or nursing women.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
* Renal insufficiency or dialysis
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
* Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) | At the end of Cycle 1 (each cycle is 28 days)
  Change of QOL after every cycle of chemotherapy assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)

SECONDARY OUTCOMES:
Rate of hand-foot skin reaction (HFSR) | At the end of Cycle 1 (each cycle is 28 days)
  Rate of HFSR after every cycle of treatment
Change of numeric rating scale (NRS) | At the end of Cycle 1 (each cycle is 28 days)
  Change of NRS and the administration of analgesic drugs after every cycle of chemotherapy. The range of NRS scale is 0-10 and higher scores mean a worse outcome.
Rate of anemia | At the end of Cycle 1 (each cycle is 28 days)
  Rate of anemia after every cycle of treatment
Overall survival (OS) | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No